CLINICAL TRIAL: NCT03080168
Title: Assessing Actigraphy-Determined Movement Variability as a Novel Objective Marker
Brief Title: The "AIM Study": Investigating Whether Actigraphy and Ideation Measures Can Promote Patient Safety
Acronym: AIM
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: MHBA-017-15S; 1I01CX001424-01 (NIH)
Record Dates: First submitted 2017-02-21; First posted 2017-03-15 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Suicidal Ideation; Suicidal Behavior; Mental Health Symptoms; Mental Health Hospitalizations
Keywords: suicidal ideation; suicidal behavior; Veterans; inpatients; Actigraphy; implicit associations; risk factors
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Actigraph: All participants will wear an Actigraph (monitoring device) for the duration of their inpatient stay.
  NOTE: In clarification, for both this section and Section 4, this devices is an FDA-regulated monitoring device, but NOT an Intervention in this study.
  Interventions: Device: Actigraph

INTERVENTIONS:
Device: Actigraph — This is NOT an intervention but a monitoring device. All participants will wear an Actigraph for the duration of their inpatient stay, as well as complete paper and computer assessments.

SUMMARY:
This is a research project looking at whether measuring movements or responses to certain questions can help predict suicidal thoughts or actions.

This project has two parts: The first part will occur while the participant is receiving hospitalized at the Bedford VA Hospital. It involves wearing a watch-like device on his/her wrist and answering questions or doing tasks to measure mood and other mental health symptoms, and suicidal thoughts.

In the second phase, the investigators will call the participant around 12 months after s/he has left the hospital. The investigators will discuss how s/he is doing and if s/he has had suicidal thoughts or made suicidal acts.

DETAILED DESCRIPTION:
As a consequence of the COVID-19 pandemic, and after consultation with the appropriate research oversight, regulatory and monitoring entities, screening and enrollment was been placed on temporary administrative hold as of 3 17 2020. As the pandemic has continued, we have reviewed our data and decided to close the study to enrollment and proceed to our analyses of findings.

RESEARCH DESIGN: A prospective cohort study of Veterans will be conducted to determine if the previously-identified specific actigraphy-based measurements highly associated with suicidal ideation in non-Veterans will predict suicidal ideation, suicidal behavior, and/or rehospitalization in Veterans.

METHODS: An analysis of Veterans admitted to the Bedford, Massachusetts VAMC acute psychiatry unit will be conducted. The primary analysis will focus upon Veterans with current suicidal ideation or recent suicidal behavior (SI/SB) who do not have a primary psychotic disorder, Alzheimer's, or Parkinson's disease, and who are not undergoing alcohol detoxification. A separate analysis will be conducted of patients undergoing alcohol detoxification, half with SI/SB and half without SI/SB. Participants will wear a small, unobtrusive, wristwatch-like actigraph on their nondominant wrist, and complete self-rated and clinician-rated assessments of suicidal ideation, as well as self-rated assessments of the severity of other psychiatric symptoms. A Resiliency Index (RI) will be calculated using nonlinear dynamic analysis of the amplitude of movements over time frames from 6 minutes - 2 hours. These time frames are the periods for which a clear structure to the movement data is evident, with patients with suicidal ideation showing less variation in amplitude than patients without suicidal ideation. If medications given for alcohol detoxification are determined to not interfere with the RI, then a secondary analysis will examine the entire sample of Veterans. One Aim will focus upon determining whether the original Resiliency Index or alternative movement data indices, such as one based on the change in the movement data over the hospitalization, predicts the presence and severity of suicidal ideation among Veteran inpatients. This aim will also examine the sensitivity and specificity of the RI for detecting the presence of any suicidal ideation, and of substantial suicidal ideation. (In non-Veterans, the RI showed a sensitivity of 72% and a specificity of 100% for detecting any suicidal ideation, and 86% and 88%, respectively, for detecting substantial ideation). In addition, the investigators may determine whether the RI predicts subsequent suicidal behavior or rehospitalization over different time periods within the original 12 month followup period, alone or combined with data about symptom severity, past history, and the present hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older and endorsing either suicidal ideation upon admission or within the last 7 days, or endorsing (or otherwise documented) suicidal behavior within the past 14 days before admission; OR
2. age 18 years or older and undergoing alcohol detoxification (including patients who qualify under #1 and are undergoing alcohol detoxification).

Exclusion Criteria:

* presence of a primary psychotic disorder [schizophrenia, schizoaffective disorder, psychosis not otherwise specified, and other psychoses] diagnosis on admission; or major depressive disorder with psychosis, or current hallucinations or ideas of reference, endorsing current psychotic thinking on the Psychosis Screen measure
* presence of a flag specifying a history of disruptive or violent behavior, or, if found during review of elements of the patient's chart prior to study enrollment, indication of a history of violent behavior towards staff, caregivers, or other patients in the patient's record, or if discussion with hospital staff indicates the potential participant's mental status is unstable enough or hostile enough to raise concerns about assaultive behavior
* Prisoner (of federal, state, or local authorities)
* Currently admitted to 78G under an involuntary commitment (e.g., "Section 12"). Specifically, no patients will be enrolled as participants who were committed to the inpatient unit involuntarily who has not chosen voluntarily to change their status to that of a voluntarily admitted patient (ie., signed a "Conditional Voluntary" form)
* Interviewer or Hospital staff-suspected or chart-documented presence of mental retardation (IQ <70) or other DSM-IV organic mental disorder (e.g., including Alzheimer's dementia)
* acute alcohol or drug intoxication or any delirium
* receiving alcohol detoxification treatment [for Primary Analysis]
* women who are pregnant
* patients undergoing detoxification for opiates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: US Veteran inpatients hospitalized for suicidal ideation, suicidal behavior, or alcohol detoxification
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
POST DISCHARGE FOLLOW-UP (COMPOSITE): CSSRS Suicidal Behaviors (self-report), Rehospitalization with Suicidal Ideation (self-report), combined with chart data re Suicidal Behavior and Rehospitalization with Suicidal Ideation | 12 months since discharge from index hospitalization
  The investigators will call some participants who are not undergoing alcohol detoxification and administer the Columbia-Suicide Severity Rating Scale to determine occurrence of all suicidal behavior (actual, interrupted, aborted, and preparatory), ask them to also self-report rehospitalization with suicidal ideation (SI), and use VA chart data as another source of information about suicidal behavior and rehospitalization.
  For those patients who we reach by phone we will use both their self-report and the information from chart review to inform this outcome, and from those patients not undergoing analysis who we don't reach, or those who are in participant groups not receiving phone calls (the participants undergoing alcohol detoxification).
  The data will then be reconciled and combined into a measure of Suicidal Behavior or rehospitalization with suicidal ideation over the 12 months since discharge.
INPATIENT: Sheehan STS scale | Last 24 hours up to assessment
  Association of Actigraph measurements with Sheehan STS Scale

SECONDARY OUTCOMES:
INPATIENT: Self-report response to Suicidal thinking diary questions re Combined Severity and Duration of suicidal thinking [Main Secondary Analysis] | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  Participants rank the Severity and Duration of their suicidal thinking on 0-10 scales each day, This outcome will look at the distribution of the interaction between the scores (e.g., multiplicative/multiplication of scores) and determine whether that simple interaction/combination will be used, log or otherwise transformed, and/or more weighting given to duration than severity, etc. This determination will be made on the spread of this data, not any information about how it correlates with actigraphy or other data gathered. This is being designated a secondary outcome simply because how the measure will be determined is not yet specified, but it is expected that this composite measure will likely have a stronger association with actigraphy and other RFs (risk factors)/predictors than simply the severity of suicidal ideation, one of the co-primary outcomes.
POST DISCHARGE FOLLOW-UP: Actual Suicidal Behavior (self-report and chart informed) [Main Secondary] | 12 months (12 months since discharge from index hospitalization)
  The investigators will use the data gathered from the CSSRS from phone interviews and chart review to determine the occurrence of Actual Suicidal Behavior in the 12 months since discharge. We will use both sources of information to assess those patients who are reached by phone and the chart review alone for those who cannot or are in the groups undergoing alcohol detoxification (who are not in the group who receive phone calls).
POST-DISCHARGE FOLLOW-UP: All Suicidal Behavior plus Rehospitalization plus Severity of Worst Suicidal Ideation (Some Intent or Some Intent or Plan) [Main Secondary] | 12 months since Discharge
  The investigators will call patients and administer CSSRS to determine, and ask about rehospitalization with SI, as well as determine information from the chart about the occurrence of these outcomes, both for patients who are reached by phone and those who cannot or are in the groups undergoing alcohol detoxification (who are not in the group who receive phone calls).
INPATIENT: Severity of Suicidal Ideation | Duration of Inpatient Stay (Daily Measures, up to 365 days [It is anticipated most subjects will provide from 2-7 days of data)
  Daily rankings of Severity of Suicidal Ideation, from the Suicidal Thinking Diary, on a scale of 0-10.
INPATIENT: Duration of Suicidal Ideation (Thinking Diary) | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  Daily rankings of Duration of Suicidal Ideation, from the Suicidal Thinking Diary, on a scale of 0-10.
INPATIENT: Duration of Suicidal Ideation (Hours/minutes) | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  Daily rankings of Duration of Suicidal Ideation, from the Sheehan Tracking Scale, in hours and minutes.
INPATIENT: Maximum Level of Suicidal Ideation per CSSRS each day | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  Maximum Level of Suicidal Ideation per CSSRS 5 Level scale (ranging from Wish to be Dead to Active Ideation with Intent and Plan).
INPATIENT: Wish to be Dead | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  Daily rankings of Wish to be Dead, from the Thinking Diary, on a 0-10 scale. [This was the outcome used in the previous actigraphy study].
INPATIENT: Combination of Maximum Level of Suicidal Ideation per CSSRS each day plus Frequency, Controllability, etc. items | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  Maximum Level of Suicidal Ideation per CSSRS 5 Level scale (ranging from Wish to be Dead to Active Ideation with Intent and Plan) combined with the items/scores in the 2nd half of the suicidal ideation assessment (frequency, controllability). Investigators will use chart and interview information for patients who can be reached by phone and interview information for those who cannot or are in the groups undergoing alcohol detoxification (who are not in the group who receive phone calls). Exact procedure for combining (e.g. simple addition) to be determined, possibly in consultation with Columbia scale staff.
Maximum severity of suicidal ideation in 12 months post-discharge (self-report, 0-10 scale) | 12 months post-discharge
  We have created our own 0-10 scale of the highest intensity of suicidal thinking a participant experienced in the 12 months post-discharge. This will be used for some of the secondary analyses of outcomes 12 months after discharge. While it is not validated, it has the advantage that, as opposed to any Yes/No events (rehospitalization, experiencing of a certain severity of suicidal thinking), that every study participant will have a value on this particular scale.

OTHER OUTCOMES:
POST-DISCHARGE FOLLOW-UP: All Suicidal Behaviors (without Rehospitalization) | 12 months post Discharge
  The investigators will call patients and administer CSSRS to determine as well as determine events from the chart, both for patients who can be reached by phone and those who cannot or are in the groups undergoing alcohol detoxification (who are not in the group who receive phone calls).
POST-DISCHARGE FOLLOW-UP: All Suicidal Behaviors, Rehospitalization with SI, and Severity of Worst Ideation involves Plan and Intent | 12 months post discharge
  The investigators will call patients and administer CSSRS to determine, and ask about rehospitalization with SI, as well as determine this information from the chart, both for patients who can be reached by phone and those who cannot or are in the groups undergoing alcohol detoxification (who are not in the group who receive phone calls).
POST-DISCHARGE FOLLOW-UP: All Suicidal Behaviors, Rehospitalization with SI, and Severity of Worst Ideation includes Method, Intent, or Plan | 12 months post discharge
  The investigators will call patients and administer CSSRS to determine, and ask about rehospitalization with SI, as well as determine the occurrence of these outcomes from the chart, both for patients who can be reached by phone and those who cannot or are in the groups undergoing alcohol detoxification (who are not in the group who receive phone calls).
INPATIENT: Nonsuicide Symptom Diary Items | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  11 items concerning psychiatric symptoms and movement/activity, on a 0-10 scale. Each will be examined individually.
INPATIENT:Sheehan STS score | 24 hours before enrollment (baseline)
  Association of the SIAT with Sheehan STS scale score for past 24 hours at baseline
INPATIENT: Combination of Sheehan Measures | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  The investigators will use Sheehan scale as an index, either: A) Weighting reach response on questions 2-6, and 8 with each question being worth 5X the previous question, and responses worth 0-4 points, depending on frequency (this will result in a scale from 0 - 4096), and/or B) a simple unweighted version which gives a score from 0 - 24 based on how frequently client endorses highest numbered item, based on specific thresholds ( a little, moderately, etc.) .
INPATIENT: Individual Sheehan Items | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  The investigators will examine the association of each Sheehan item, questions 2-6 and 8 with the actigraph and other predictors.
INPATIENT: CSSRS Duration Item | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  Suicidal Ideation Item on CSSRS.
INPATIENT: CSSRS at baseline | 1-2 weeks pre-enrollment
  Association of the SIAT with Level of Suicidal thinking (0-5) on Columbia Scale (CSSRS) at baseline (over last week for SI, last 2 weeks for SB)
INPATIENT: CSSRS Frequency Item | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  Suicidal Ideation Item on CSSRS.
INPATIENT: Duration of Suicidal Thinking | 24 hours pre-enrollment
  Association of the SIAT with Duration of Suicidal Thinking (0-10) Today
INPATIENT: CSSRS Frequency/Duration Item combination | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  The investigators will use some combination of the Frequency and Duration item (either simple addition or multiplication, or some other combination, taking into account as frequency increases the maximum duration must at some point decrease).
INPATIENT: PHQ-9 score Item 9 (0-3) | 2 weeks pre-enrollment (baseline)
  Association of the SIAT with PHQ-9 score Item 9 (Frequency for last 2 weeks, including better off dead) for last 2 weeks
INPATIENT: CSSRS Controllability Item | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  Suicidal Ideation Item on CSSRS.
INPATIENT: CSSRS Deterrents Item | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  Although this will be analyzed, it is not expected this will correlate as much with actigraphy or other predictors than other CSSRS items.
INPATIENT: CSSRS Reasons Item | Duration of Inpatient Stay (Daily Measures, up to 365 days)
  Although this will be analyzed, it is not expected this will correlate as much with actigraphy or other predictors than other CSSRS items.
POST-DISCHARGE FOLLOW-UP: Actual Suicidal Behavior with Lethality of 1+ on CSSRS | 12 months post-discharge
  Suicidal behavior, only counting behaviors of a certain level of lethality.
INPATIENT:Sheehan Tracking System | 24 hours pre-enrollment (baseline)
  Association of the SIAT with Sheehan STS scale score for past 24 hours at baseline.
INPATIENT: Change in Severity or Duration of Suicidal Thinking or the Composite Measure | Inpatient (Daily Measures, Days 1 and 2 combined versus last 1, 2, or 3 days [longest period up to 3 days that does not overlap with days 1&2)
  For analyses examining CHANGE in the Actigraph index, or CHANGE in the Actigraph index plus change in some of the other predictors, the investigators will examine an outcome involving Change in Suicidal Thinking (probably the measure most predictive in the earlier analyses of the level of the index/predictors and the severity/duration of suicidal thinking).
POST-DISCHARGE FOLLOW-UP: Actual Suicidal Behavior with Lethality 2+ on CSSRS | 12 months (post-discharge
  Suicidal behavior, only counting behaviors of a certain level of lethality.
INPATIENT: Sheehan Tracking System | 24 hours pre-enrollment (baseline)
  Association of the Sheehan STS scale score for the 24 hours prior to enrollment (baseline) with the Actigraph movement index (called to this point the Vulnerability Index, but we may invert and call it the Resiliency index), for days 1-3 of the study.
INPATIENT: Sheehan Tracking System | 24 hours pre-enrollment (baseline)
  Association of the Sheehan STS scale score for the 24 hours prior to enrollment (baseline) with a modified (shorter time-frame) version of the Actigraph movement index (called to this point the Vulnerability Index, but we may invert the index and call the Resiliency Index), for day 1 of the study, day 1 and 2 of the study combined, or both.
INPATIENT: CSSRS at baseline | 1-2 weeks prior to enrollment (baseline)
  Association of the Level of Suicidal thinking (0-5) on Columbia Scale (CSSRS) at baseline (over last week for SI, last 2 weeks for SB) with the Actigraph movement index (called to this point the Vulnerability Index, but we may invert the index and call it the Resliency index), for days 1-3 of the study.
INPATIENT: CSSRS at baseline | 1-2 weeks prior to enrollment (baseline)
  Association of the Level of Suicidal thinking (0-5) on Columbia Scale (CSSRS) at baseline (over last week for SI, last 2 weeks for SB) with a modified (shorter time-frame) version of the Actigraph movement index (called to this point the Vulnerability Index, but we may invert and call the Resiliency Index, for day 1 of the study, day 1 and 2 of the study combined, or both.
INPATIENT: Duration of Suicidal Thinking | Day of enrollment but for the hours prior to enrollment (baseline)
  Association of the Duration of Suicidal Thinking (0-10) Today item of the Thinking Diary at baseline with the Actigraph movement index (called to this point the Vulnerability Index, but we may invert the index and call it the Resiliency index), for days 1-3 of the study.
INPATIENT: Duration of Suicidal Thinking | Day of enrollment but for the hours prior to enrollment (baseline)
  Association of the Duration of Suicidal Thinking (0-10) Today item of the Thinking Diary at baseline with a modified (shorter time-frame) version of the Actigraph movement index (called to this point the Vulnerability Index, but we may invert and call the Resiliency Index, for day 1 of the study, day 1 and 2 of the study combined, or both.
INPATIENT: PHQ-9 Item 9 Score (0-3) | 2 weeks prior to enrollment (baseline)
  Association of the PHQ-9 score for Item 9 (Frequency over the last 2 weeks of thoughts of self-harm, or thoughts would be better off dead) with the Actigraph movement index (called to this point the Vulnerability Index, but we may invert the index and call it the Resiliency index), for days 1-3 of the study.
INPATIENT: PHQ-9 Item 9 Score (0-3) | 2 weeks prior to enrollment (baseline)
  Association of the PHQ-9 score for Item 9 (Frequency over the last 2 weeks of thoughts of self-harm, or thoughts would be better off dead) with a modified (shorter time-frame) version of the Actigraph movement index (called to this point the Vulnerability Index, but we may invert and call the Resiliency Index, for day 1 of the study, day 1 and 2 of the study combined, or both.
Wish to be Dead (0-10) scale at baseline | Baseline (that day)
  We will derive the Pearson correlation coefficient between the S-IAT d score at Baseline and their reported Wish to be Dead that day at baseline (ie., not considering any data from the subsequent hospitalization). This is being performed as pilot analysis to support a grant application.
Wish to be Dead (0-10) scale at baseline | Baseline (that day)
  We will derive the Pearson correlation coefficient between the Actigraphy Vulnerability Index (also known as the Resiliency Index if the scores are inverted) their reported Wish to be Dead that day at baseline (ie., not considering any data from the subsequent hospitalization). This is being performed as pilot analysis to support a grant application.

CONTACTS AND LOCATIONS:
Overall Officials: Eric G. Smith, MD PhD MPH, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA
Locations (1):
- Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT03080168/ICF_000.pdf